CLINICAL TRIAL: NCT01965379
Title: Effect of Restriction of Foods Containing Phosphorus Additives on the Phosphatemia of Patients With End-stage Renal Disease.
Brief Title: Effect of Restriction of Foods Containing Phosphorus Additives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Margareth Lage Leite de Fornasari, PHD student, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Fornasari01
Record Dates: First submitted 2013-10-09; First posted 2013-10-18 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: End-stage Renal Disease; Hyperphosphatemia
Keywords: Dialysis; Phosphorus; Diet
MeSH Terms: conditions — Kidney Failure, Chronic; Hyperphosphatemia | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): Restriction on food containing phosphorus additives.
  Interventions: Other: Restriction on food containing phosphorus additives
- Control (Placebo Comparator): Standard care.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Restriction on food containing phosphorus additives — The substitution of foods containing phosphorus additives for others with the same nutritional value for each individual of the study.
  Arms: Intervention
Other: Standard care — The control group mantained the usual renal diet oriented prior to the study with a booklet.
  Arms: Control

SUMMARY:
Hyperphosphatemia is related to the increase in morbidity and mortality. There is greater risk for cardiovascular disease, atherosclerotic disease, secondary hyperparathyroidism, and bone disease .

The serum phosphorus level can be controlled by a combination of factors, such as: reduction of ingestion, reduction of intestinal absorption with chelating agents and increase in elimination by dialysis.

The purpose of this study is to evaluate the effect of dietary intervention consisting of the restriction of industrialized foods with phosphorus additives in chronic kidney disease patients treated with hemodialysis.

DETAILED DESCRIPTION:
The consumption of foods which contain phosphorus by patients on hemodialysis should be monitored in order to reflect the current reality, due to the increase in ingestion of industrialized foods rich in phosphorus additives. Data from studies performed in the USA shows a reduction in phosphatemia with nutritional orientation to reduce foods containing additives from restaurants in the region of the study . In another study, also conducted in the USA, the researchers evaluated the phosphorus content and presence of additives in appetizers and side orders served at fast food restaurants in Cleveland. The results showed that of the appetizers, 52% were accepted by the traditional criteria for the renal diet (low content of sodium, potassium and organic or natural phosphorus), but only 16% were also free of phosphorus additives; of the side orders, 23% were accepted by the traditional criteria and 17% were exempt of phosphorus additives. Thus, only a small proportion of appetizers and side orders served at fast food restaurants were compatible with the renal diet. Considering that alimentary phosphorus has an important role in the control of phosphatemia, there is a lack of studies which evaluates the effect of foods containing phosphorus additives on phosphatemia and which, at the same time, evaluated the alimentary ingestion and the nutritional state of the chronic kidney disease patients treated with hemodialysis.

Can the elimination of foods containing phosphorus additives and their substitution for foods without additives reduce phosphatemia without altering the nutritional state of hyperphosphatemic patients on hemodialysis?

ELIGIBILITY:
Inclusion Criteria:

* males or female ≥ 18 years of age
* Chronic kidney disease in stage 5, on hemodialysis for at least 6 months
* Serum phosphorus (P) greater than 5.5 mg/dL persistent in 3 previous months
* Preserved cognitive capacity and able to read and write
* Signed informed written consent

Exclusion Criteria:

* Use of enteral or parenteral therapy
* Presence of physical or cognitive limitation
* Malabsorption diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change the serum levels of phosphorus to acceptable levels ( under 5.5 mg per dL) | 90 days

SECONDARY OUTCOMES:
Protein intake at baseline and final. | 90 days
Energy intake at baseline and at the final. | 90 days
Triceps skinfold at baseline and final. | 90 days
Body mass index at baseline and final | 90 days
Arm muscle area at baseline and final | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Yvoty AS Sens, PHD, Study Chair — Faculdade de Ciências Médicas da Santa Casa de São Paulo; Margareth LL Fornasari, RD, Principal Investigator — Faculdade de Ciências Médicas da Santa Casa de São Paulo
Locations (1):
- Faculdade de Ciências Médicas da Santa Casa de São Paulo, São Paulo, São Paulo, Brazil